CLINICAL TRIAL: NCT00212550
Title: Evaluation of the Practice of Three Morning Sputa on Separate Days for Diagnosis of Mtb
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 9250-04B
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Pulmonary TB
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TB diagnosis
  Interventions: Procedure: Obtain standard three daily sputum samples vs. three samples on the first day for the diagnosis of pulmonary TB.

INTERVENTIONS:
Procedure: Obtain standard three daily sputum samples vs. three samples on the first day for the diagnosis of pulmonary TB. — Sputum induction

SUMMARY:
Obtain sputum smears within one day to rule out TB

ELIGIBILITY:
Inclusion Criteria:

* All subjects admitted to Bellevue Hospital for evaluation of possible TB

Exclusion Criteria:

* Unable to produce spontaneous or induced sputum

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TB patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2006-01; Primary Completion 2010-02 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rany Condos, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU School of Medicine Division of Pulmonary and Critical Care, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided